CLINICAL TRIAL: NCT01378325
Title: Crystalloid Coload Combined With Variable Rate Phenylephrine Infusion for Prevention of Hypotension During Spinal Anesthesia for Elective Cesarean Delivery vs Crystalloid Coload Alone
Brief Title: Variable Rate Phenylephrine Infusion for Prevention of Spinal-induced Hypotension for Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sahar Sayyid, anesthesia, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANES.SS.10
Record Dates: First submitted 2011-06-10; First posted 2011-06-22 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Anesthetic Complication Spinal
Keywords: spinal; cesarean delivery; phenylephrine; hypotension
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylephrine (Experimental): PHenylephrine infusion started at 0.75 microgram per kg per mL started at spinal injection till delivery
  Interventions: Drug: Phenylephrine
- Saline (Placebo Comparator): Prophylactic variable rate of saline infusion where we adjusted the pump at a starting rate of 0.75 µg/kg/min, equivalent to 0.0075 mL/kg/min of saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Phenylephrine — Prophylactic variable rate of phenylephrine infusion started at 0.75 µg/kg/min vs saline
  Other Names: Neosynephrine
  Arms: Phenylephrine
Drug: saline — Prophylactic variable rate of saline infusion where we adjusted the pump at a starting rate of 0.75 µg/kg/min, equivalent to 0.0075 mL/kg/min of saline
  Arms: Saline

SUMMARY:
Rapid administration of crystalloid immediately after induction of spinal anesthesia (coload) to be more effective in terms of managing hypotension as compared to administering crystalloid before spinal anesthesia (preload).

Phenylehrine infusion is a safe and effective way to reduce incidence and frequency of hypotension during SA for cesarean delivery. Hypotension was virtually eliminated by use of high-dose prophylactic phenylephrine infusion at a rate of 100 µg/min and rapid crystalloid coload up to two liters (administration at the time of SA). However, incidence of reactive hypertension was frequent up to 47% with decrease in maternal heart rate (HR). This may raise concern in patients in whom increase of blood pressure may be detrimental, like chronic hypertension and in the presence of a compromised uteroplacental blood flow. A recent study found that infusing phenylephrine at a fixed rate of 75 and 100 ug/min is associated with more episodes of hypertension than placebo or the lower infusion rates of 25 and 50 ug/min respectively. However, there was no reduction in the number of physician interventions (phenylephrine boluses and stopping the infusion) needed to maintain maternal systolic blood pressure within 20% of baseline among all groups. Prophylactic fixed rate infusions may have limited application in clinical practice, and a variable rate (i.e. modifying the rate according to hemodynamics) has been advocated. The bolus administration of phenylephrine to treat hypotension is still commonly used, but requests multiple interventions from the anesthesiologists and is time consuming.

Eighty patients scheduled for cesarean delivery under spinal anesthesia will be assigned to one of two groups. Immediately after spinal injection, rapid crystalloid colaod of lactated Ringer of 15 mL/kg over a period of 10-15 min will be initiated. Patients in Group I will receive infusion of normal saline (placebo) and patients in group II variable infusion rate of phenylephrine started at 0.75 ug/kg (close to the dose of 50 ug/min recommended for fixed infusion rate). The number of interventions needed to maintain maternal systolic blood pressure within 20% of baseline, hemodynamic performance, intraoperative nausea and vomiting, and umbilical cord blood gases will be compared between the two groups.

We will define a reliable and safe method to ensure maternal hemodynamic stability during spinal anesthesia for cesarean delivery with the least physician interference.

ELIGIBILITY:
Inclusion Criteria:

* Parturients beyond 37 weeks gestation
* ASA І or ІІ

Exclusion Criteria:

* pregnancy-induced hypertension
* chronic hypertension
* multiple pregnancy
* fetal compromise
* diabetes mellitus
* polyhydramnios
* body weight >100 kg
* major systemic disease
* anemia (hemoglobin concentration<10 g/dl)
* clotting diathesis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: crystalloid coload with lactated Ringer solution combined with prophylactic variable rate of saline infusion where we adjusted the pump at a starting rate of 0.75 µg/kg/min, equivalent to 0.0075 mL/kg/min of saline
Period: Overall Study
Arm/Group | Phenylephrine | Saline
Started | 40 | 40
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: with β of 0.2 and α of 0.05 and two-sided test for comparing two means (http://www.stat.ubc.ca/~rollin/stats/ssize/n2.html), the calculated number of patients was 37 in each group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Phenylephrine | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (5) | 32.5 (5) | 33 (5)
Sex/Gender, Customized [Number; unit: participants] — Gender, female
  participants
    Number of Female Participants | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Number of Physician Interventions Needed to Maintain Maternal Blood Pressure After Spinal Anesthesia Within 20% of Baseline and to Treat Bradycardia During Cesarean Delivery.
Description: Physician interventions are triggered by hemodynamic changes more than 20% of baseline. The intervention can be one or more of the following:
  * stopping the phenylephrine infusion
  * changing the rate of phenylephrine infusion
  * rescue intravenous bolus of phenylephrine (100 µg) for hypotension
  * rescue intravenous bolus of atropine (0.4 mg) for bradycardia
Time Frame: Patients will be followed up throughout the Cesarean delivery (average of 1.5 hours).
Measure: Median (Full Range); unit: number of interventions
Arm/Group | Phenylephrine | Saline
Number analyzed (Participants) | 40 | 39
number of interventions | 0 [0 to 6] | 3 [0 to 9]

ADVERSE EVENTS:
Arm/Group | Saline | Phenylephrine
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/39 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No